CLINICAL TRIAL: NCT05783050
Title: Comparison of Wei Nasal Jet Tube and Nasal Cannula Oxygen Support Methods in Sedated Gastrointestinal Endoscopy Patients: A Prospective, Randomized Controlled Study
Brief Title: Wei Nasal Jet Tube vs Nasal Cannula Oxygen Support in Gastrointestinal Endoscopy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, İsmail SÜMER, Principal Investigator, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Ismail04
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Supraglottic Airway Obstruction; Airway Complication of Anesthesia; Airway Obstruction; Anesthesia Complication; Bronchospasm; Nasal Bleeding; Oxygen Deficiency
Keywords: Wei Nasal Jet Tube; Airway Complication; Nasal Cannula Oxygen Support; Gastrointestinal Endoscopy; sedation
MeSH Terms: conditions — Airway Obstruction; Bronchial Spasm; Epistaxis; Hypoxia

STUDY DESIGN:
Who Masked: Participant
Masking Description: computer-assisted randomization method
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wei Nasal Jet Tube Group (Group W) (Active Comparator): After induction of anesthesia, the Wei Nasal Jet Tube was placed in the patients.
  Interventions: Device: Wei Nasal Jet Tube
- Nasal Cannula Oxygen Support Group (Group N) (Active Comparator): After the induction of anesthesia, the Nasal Cannula Oxygen Cannula was placed in the patients.
  Interventions: Device: Nasal Cannula Oxygen Support

INTERVENTIONS:
Device: Wei Nasal Jet Tube — The purpose of this procedure is to provide safe oxygenation and ventilation. While providing oxygen support, nasal cannula, classical oxygen mask can be used, as well as new generation oxygenation devices.
  Arms: Wei Nasal Jet Tube Group (Group W)
Device: Nasal Cannula Oxygen Support — The purpose of this procedure is to provide safe oxygenation and ventilation. While providing oxygen support, nasal cannula, classical oxygen mask can be used, as well as new generation oxygenation devices.
  Arms: Nasal Cannula Oxygen Support Group (Group N)

SUMMARY:
Sedoanalgesia is applied to patients during gastrointestinal endoscopy. Sedoanalgesia may cause respiratory depression and hypoxia in patients. During these procedures, patients should be given oxygen support to reduce the incidence of hypoxia.This study aimed to compare the efficacy and procedural performance of two different airway devices (Wei Nasal Jet Tube vs Nasal Cannula Oxygen Support) in Gastrointestinal Endoscopy

DETAILED DESCRIPTION:
Gastrointestinal endoscopy is performed as standard for the diagnosis of many gastrointestinal diseases. During gastrointestinal endoscopy, sedoanalgesia is applied to relieve patients' pain and increase patient comfort. Anesthetic drugs used for sedoanalgesia may cause respiratory depression and hypoxia in patients. Hypoxia resulting from hypoventilation in patients is responsible for many events, including coronary ischemia. During these procedures, patients should be given oxygen support to reduce the incidence of hypoxia. The purpose of this procedure is to provide safe oxygenation and ventilation. While providing oxygen support, nasal cannula, classical oxygen mask can be used, as well as new generation oxygenation devices. Our study will show us which method is more beneficial in preventing hypoxia and other side effects, providing comfort for the doctor performing the procedure and for the patient undergoing the procedure. This study aimed to compare the efficacy and procedural performance of two different airway devices (Wei Nasal Jet Tube vs Nasal Cannula Oxygen Support) in Gastrointestinal Endoscopy

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing gastrointestinal endoscopy
* ASA Physical Status 1-2
* Body mass index 18.5 - 35 kg/m2

Exclusion Criteria:

* High risk of pulmonary aspiration

  * Pregnancy
  * Anesthesic drug allergies
  * Difficult airway or facial deformities
  * Height <155 cm
  * Alcohol or narcotic drug usage
  * Restrictive or obstructive pulmonary diseases
  * Hepatic cardiac or renal failure
  * Neurologic or cognitive deficiencies.
  * Previous cervical surgery or cervical radiotherapy
  * Previous esophagus surgery
  * Psychotic problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Hypoxia incidence | Intra-operative; after device insertion
  Hypoxia is defined as SpO2 <92% at any time.

SECONDARY OUTCOMES:
Airway assist maneuver required | Intra-operative; after device insertion
  When the SpO2 value is below 90-92%, airway support maneuvers will be performed
Procedure failure incidence | Intra-operative; after device insertion
  The development of severe hypotension (MAP <55 mmHG), bradycardia ( HR< 45 bpm) and prolonged deep hypoxia(>60 sec SpO2<92%) during procedure

CONTACTS AND LOCATIONS:
Overall Officials: ISMAIL SUMER, MD, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)